CLINICAL TRIAL: NCT03380559
Title: A Phase III Randomized Double-blind Study to Evaluate Efficacy of Botulinum Toxin for Treating Epicondylitis
Brief Title: A Phase III Study to Evaluate Efficacy of Botulinum Toxin for Treating Epicondylitis
Acronym: EPITOX
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P160926J; 2017-001709-33 (EudraCT Number)
Record Dates: First submitted 2017-12-11; First posted 2017-12-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Epicondylitis
Keywords: Epicondylitis; Botulinum toxin; Corticoid
MeSH Terms: interventions — Injections; Botulinum Toxins; Adrenal Cortex Hormones

STUDY DESIGN:
Intervention Model Description: Ratio 1:1:1
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A : Association (botulinum toxin + corticoid) (Experimental)
  Interventions: Drug: Injection, botulinum toxin + corticoid
- Group C : placebo of toxin + corticoid : (Placebo Comparator)
  Interventions: Drug: Injection, placebo of toxin + corticoid
- Group T : botulinum toxin + placebo corticoid (Active Comparator)
  Interventions: Drug: Injection, botulinum toxin + placebo corticoid

INTERVENTIONS:
Drug: Injection, botulinum toxin + corticoid — * Intramuscular injection of botulinum toxin (Xeomin® 50 U) under ultrasound control
  * Subcutaneous injection (lateral epicondylitis side) of corticoid (2 ml of Hydrocortancyl® 2,5 %)
  Arms: Group A : Association (botulinum toxin + corticoid)
Drug: Injection, placebo of toxin + corticoid — * Intramuscular injection of placebo botulinum toxin (2 ml) under ultrasound control
  * Subcutaneous injection (lateral epicondylitis side) of corticoid (2 ml of Hydrocortancyl® 2,5 %)
  Arms: Group C : placebo of toxin + corticoid :
Drug: Injection, botulinum toxin + placebo corticoid — * Intramuscular injection of botulinum toxin (Xeomin® 50 U) under ultrasound control
  * Subcutaneous injection (lateral epicondylitis side) of placebo of corticoid (2 ml of physiological saline solution NaCL 0.9 %)
  Arms: Group T : botulinum toxin + placebo corticoid

SUMMARY:
The study aims to demonstrate that intramuscular injection of botulinum toxin with a paralyzing dose coupled with subcutaneous injection of corticoid has greater efficacy than corticoid injection only or toxin injection only for treating lateral epicondylitis in reducing pain at 6 months.

As secondary objectives, the study aims to

* demonstrate improvement of quality of patient's life and positive effect on their resuming to professional activities or sportive activities.
* evaluate tolerance of treatment by grip strength measurement and adverse event collection.

DETAILED DESCRIPTION:
This is a prospective multicenter phase IIIb randomized double-blind placebo-controlled study, to compare efficacy and tolerance of 3 groups of treatments for epicondylitis.

All patients will be randomized in 3 following parallel treatment groups:

Group A : botulinum toxin + corticoid

Group C : placebo of toxin + corticoid

Group T : botulinum toxin + placebo corticoid

The study will be performed in 4 centers in France, targetting 150 patients. The follow-up of each patient will last 6 months after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged between 18 and 60 years;
* Physical disability or not;
* Unilateral lateral epicondylitis more than 3 months, recurrent or not, no response to at least one standard treatment such as: local injection of corticoid, physiotherapy, rest, NSAIDs per os;
* Signed consent obtained;
* Covered by health insurance.

Exclusion Criteria:

* Central nervous system disorders result in spasticity in epicondylitis limb;
* History of severe psychiatric disorder;
* History of myasthenia gravis;
* Pregnant or breastfeeding woman;
* Unable to understand or respond to questions;
* Contraindication to botulinum toxin or corticoid;
* Treatment with botulinum toxin 3 months prior to baseline;
* Anticoagulant theraphy;
* Difficult to follow-up in the study;
* Patient under guardianship, or deprived of liberty by a judicial order.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2019-04-19 (Actual); Primary Completion 2021-07-07 (Actual); Study Completion 2021-08-19 (Actual)

PRIMARY OUTCOMES:
Variation of pain intensity between injection of treatment and 6 months after injection | At the moment of injection
  Evaluate the variation of muscle pain intensity in wrist extensor contractions between the moment of injection and the end of the 6th month with the Visual Analogue Scale (VAS).
Variation of pain intensity between injection of treatment and 6 months after injection | 6 months after injection
  Evaluate the variation of muscle pain intensity in wrist extensor contractions between the moment of injection and the end of the 6th month with the VAS.

SECONDARY OUTCOMES:
Spontaneous pain intensity at rest | Before injection, 3 months after injection and 6 months after injection
  Evaluate pain intensity at rest with the VAS.
Pain intensity of motion of wrist flexion | Before injection, 3 months after injection and 6 months after injection
  Evaluate pain intensity of motion of wrist flexion with the VAS.
Pain intensity at proximal insertion palpation on epicondylitis muscle | Before injection, 3 months after injection and 6 months after injection
  Evaluate pain intensity at proximal insertion palpation on epicondylitis muscle. The palpation will be under ultrasound control.
Number of days of sick leave | 6 months after injection
  Number of days of sick leave will be noted and collected
The percentage of patients returning to professional activity or sportive activity | 6 months after injection
Measurement of prehensile grasp capabilities by a force | At baseline, 3 months after injection, 6 months after injection
  The force will be measured by Jamar Hydraulic hand dynamometer.
Functional outcome after injection | At baseline, 3 months after injection, 6 months after injection
  Outcome will be evaluated by questionnaire Patient Rated Tennis Elbow Evaluation
Anxiety and depression tests | At baseline, 3 months after injection, 6 months after injection
  Hospital Anxiety and Depression scale will be used
Frequence and gravity of adverse events | At baseline, 3 months after injection, 6 months after injection
  Adverse events will be collected and their severity will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: François Genêt, MD, PhD, Study Chair — Service de Médecine Physique et de Réadaptation Hôpital Raymond Poincaré
Locations (1):
- Service de Médecine Physique et de Réadaptation, Hôpital Raymond Poincaré, Garches, Hauts-de-Seine, France

IPD SHARING:
Plan to Share IPD: No